CLINICAL TRIAL: NCT06296797
Title: Disseminating PCOR Findings to Reduce Racial Disparities in Surgical Sterilization
Brief Title: Patient-centered Information on Permanent Contraception
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Essential Access Health (Other); Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 5R18HS029432-02 (AHRQ); R18HS029432 (AHRQ)
Record Dates: First submitted 2024-01-02; First posted 2024-03-06 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Contraception; Reproductive Behavior; Contraception Behavior
Keywords: tubal sterilization; permanent contraception; intrauterine device; contraceptive implant; vasectomy
MeSH Terms: conditions — Reproductive Behavior; Contraception Behavior

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comparative information on tubal sterilization and other long-acting contraceptives (Experimental): A new website comparing tubal sterilization to vasectomy and long-acting reversible contraceptives
  Interventions: Behavioral: Advancing Access Website
- Information on tubal sterilization (Active Comparator): Participants will be shown an existing web page developed by Planned Parenthood for people considering tubal sterilization
  Interventions: Behavioral: Control arm: Existing educational website

INTERVENTIONS:
Behavioral: Control arm: Existing educational website — Information about tubal sterilization currently provided on the Planned Parenthood website
  Arms: Information on tubal sterilization
Behavioral: Advancing Access Website — A website comparing tubal sterilization to long-acting reversible contraceptives informed by recent patient centered outcomes research.
  Other Names: Comparisons of tubal sterilization to long-acting reversible contraceptives
  Arms: Comparative information on tubal sterilization and other long-acting contraceptives

SUMMARY:
The goal of this study is to understand whether providing information to women with a strong desire to avoid future pregnancy about how tubal sterilization compares to long-acting reversible contraceptives improves perceived access to available contraceptives.

Participants will:

* Complete a baseline survey
* Receive access to web-based educational resources
* Complete a brief follow up survey immediately after exploring these web-based resources
* Complete a follow-up survey 3 months after enrolling

The investigators will compare outcomes among participants provided with access to a new website (intervention) summarizing recent patient-centered outcomes research (PCOR) comparing interval laparoscopic tubal sterilization and long-acting reversible contraception (LARC) to control participants provided with access to the existing Planned Parenthood website on tubal sterilization.

DETAILED DESCRIPTION:
This study evaluates the potential benefits of web-based resources to prepare patients considering tubal sterilization to effectively communicate their personal values and priorities to their clinicians, informed by recent patient centered outcomes research (PCOR) comparing interval tubal sterilization to long-acting reversible contraceptives. The investigators hypothesize that patients provided with information on the comparative safety and effectiveness of all available long acting contraceptives will be more likely to obtain contraceptive care that aligns with their personal preferences. The short-term goal of this work is to support patient-centered contraceptive care by increasing knowledge of and perceived access to all available long acting contraceptives among those who wish to avoid future pregnancy. The long-term goal of this work is to increase the proportion of women who are using a method of contraception that aligns with their personal preferences, reduce the proportion of women who regret having undergone a permanent contraceptive procedure, and reduce racial disparities in surgical sterilization.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported fertility
* Have a strong desire to avoid future pregnancy
* Speak English or Spanish

Exclusion Criteria:

* Current pregnancy
* The inability to speak English or Spanish
* Prior tubal sterilization or "Essure" procedure
* Menopause
* Infertility
* Hysterectomy

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 650 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Perceived Access to Long Acting Contraceptives | Immediately after introduction to website and at 3 months follow-up
  A 9-item, multi-dimensional measure assessing awareness, availability, accessibility, affordability, and acceptability of contraceptive options including tubal sterilization, vasectomy, the subdermal implant, hormonal intrauterine device, and hormone-free intrauterine device. A summative score ranging from 0 to 48 points will be calculated for each participant at baseline and follow up. Investigators hypothesize there will be greater improvements from baseline to follow up in the intervention than control arm.

SECONDARY OUTCOMES:
Person-Centered Contraceptive Counseling Measure | 3 month follow-up
  4-items including: Letting me say what mattered to me about my birth control, Taking my preferences about my birth control seriously, Giving me enough information to make the best decision about my birth control method, Respecting me as a person, with responses range from 1 ("Strongly Disagree") to 5 ("Strongly Agree"). Investigators hypothesize there will be greater improvements from baseline in the intervention than control arm.
Consumer Assessment of Healthcare Providers and Systems | 3 months follow-up
  Response options on a 10-point Likert scale, ranging from poor (0) to excellent (10).
  Investigators hypothesize there will be greater improvements from baseline in the intervention than control arm.
Patients' Perceived Efficacy in Patient-Physician Interactions (PEPPI) | immediately after introduction to website and 3 months follow-up
  To create a score on the 5 item contraceptive "PEPPI scale" ranging from 5 (lowest possible score) to 25 (representing highest patient-perceived self-efficacy), each item begins with "How confident are participants in their ability to… ", and subjects respond to each question on a scale of 1 to 5, with 5 representing "very confident," and 1 representing "not at all confident" Investigators hypothesize there will be greater improvements from baseline to follow up in the intervention than control arm.
Knowledge of Long-Acting Contraceptives | Immediately after introduction to website and at 3 month follow-up
  10 items adapted from the previously used Tubal Sterilization Knowledge Questionnaire items developed by Hall et al. Answers will be coded as correct vs. incorrect (with "Don't Know" being coded as an incorrect response) to create a knowledge score. Investigators will calculate change in knowledge scores on follow up surveys compared to baseline. Investigators hypothesize there will be greater improvements from baseline in the intervention than control arm.
Use of preferred method of contraception | 3 month follow-up
  3 items detailed in prior publication (PUBMED Number: 27710196)
Would recommend website to a friend | Immediately after introduction to website, and at 3 month follow up
  5 items designed to evaluate usability of website and recommendations to friends. E.g., "Using a scale of 0 (not at all) to 10 (extremely likely), participants will indicate how likely they are to recommend this website to a friend who is considering getting her tubes tied? (0-10)"

OTHER OUTCOMES:
Suggestions for how to improve web-based resources for people considering permanent contraception. | immediately following introduction to website and at 3 months follow-up
  Open-ended question regarding ease-of-use and helpfulness of the web-based program. These responses will provide ongoing information to help guide future adaptations and dissemination.

CONTACTS AND LOCATIONS:
Overall Officials: Eleanor Schwarz, MD, MS, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schwarz EB, Lewis CA, Dove MS, Murphy E, Zuckerman D, Nunez-Eddy C, Tancredi DJ, McDonald-Mosley R, Sonalkar S, Hathaway M, Gariepy AM. Comparative Effectiveness and Safety of Intrauterine Contraception and Tubal Ligation. J Gen Intern Med. 2022 Dec;37(16):4168-4175. doi: 10.1007/s11606-022-07433-4. Epub 2022 Feb 23. PMID 35194746